CLINICAL TRIAL: NCT07262086
Title: Clinical Evaluation of Wear Resistance and Bioactivity of Self Cured Bioactive Resin Composite
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1016/2025; 1016/2025 (Other: suez canal university)
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-11

CONDITIONS: Dental Caries; Class II Dental Caries
Keywords: dental caries; wear resistance; bioactive resin composite
MeSH Terms: conditions — Dental Caries | interventions — Resins, Plant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Light cured nanohybrid RBC restorations (Sham Comparator): Conventional nanohybrid composite placement for Class II restorations
  Interventions: Procedure: Resins, Composite nanohybrid
- "Self-cured Bioactive Resin Composite." (Experimental): Self-cured bioactive composite placement for Class II restorations
  Interventions: Procedure: Resins, Composite bioactive

INTERVENTIONS:
Procedure: Resins, Composite nanohybrid — Placement of light-cured nanohybrid resin composite for Class II restorations, following manufacturer's instructions
  Other Names: conventional nanohybrid resin composite
  Arms: Light cured nanohybrid RBC restorations
Procedure: Resins, Composite bioactive — Placement of self-cured bioactive resin composite for Class II restorations, following manufacturer's instructions
  Other Names: bioactive composite
  Arms: "Self-cured Bioactive Resin Composite."

SUMMARY:
Introduction:

Resin-based composites (RBCs) have become the gold standard in restorative dentistry due to their superior aesthetics, adhesion, and minimally invasive application. However, wear remains a critical drawback, compromising their longevity and clinical performance. Various techniques have been suggested to measure the clinical performance of (RBCs). Recent advancements in digital dentistry, such as intraoral scanning, offer a more precise and efficient approach for quantitative wear assessment.

Aim:

This study aims to evaluate wear resistance and bioactivity of self cured bioactive resin composite vs nanhybrid resin composite.

Methodology:

Twelve healthy patients with 24 carious molar teeth will be selected where each patient should have two oclusso- mesial cavities. Standardized oclusso- mesial cavities will be prepared for all the selected teeth, for each patient the first tooth will be restored with conventional nanohybrid RBC (M1). Meanwhile, the second tooth will be restored by self-cure bioactive RBC (M2). Then, wear resistance will be evaluated by intraoral scanner immediately after restoration (T0), six months later (T1), after 12 months (T2), 18 months (T3) and 24 months (T4). Software analysis will be done by superimposing the 3D digital impression and evaluate the restoration wear by calculating the 3D volume loss.

Also, bioactivity of the restoration will be measured by measuring the mineral density beneath the restoration. Digital radiographic images will be taken for the restoration by parallel technique and grey scale of the pixels under restoration will be measured by software immediately after restoration (D0), one month later (D1) and after 3 months (D2).

DETAILED DESCRIPTION:
II- 1 Study Setting:

A randomized controlled double-blinded clinical trial will be conducted where both patient and examiners will be blinded to the group assignment. Patients of age group 21-45 years will be selected where each patient should have two oclusso- mesial cavities. Patients will be recruited from the outpatient clinic of Conservative Dentistry department in the Faculty of Dentistry, Suez Canal University. During the initial examination, the purpose and the method of the research will be explained to the patients and a written informed consent will be assigned by each individual.

II-2 Sample Selection:

Patients participating in this study will be selected according to the following eligibility criteria:

II-2-a Inclusion Criteria:

1. Patients with vital two molar teeth with compound class II deep carious lesions.
2. Both males and females will be included.
3. Patients with good general health.
4. Patients with good oral hygiene.
5. Co-operative patients.
6. Absence of spontaneous pain, mobility or tenderness on percussion.
7. Radiographically: no internal or external resorption, no periapical or furcation radiolucency and no widening of the periodontal ligament space.

II-2-b Exclusion Criteria:

1. Patients with systemic decease.
2. Patients with severe or chronic periodontitis.
3. Patients have allergy to the materials used in this trial.
4. Nonfunctioning teeth.
5. Teeth with any pathologic pulpal changes.
6. Teeth with previous restorations.
7. Teeth with surface loss due to non carious lesions. All patients who will attend the clinic will receive the proposed treatment protocols. However, only those who will meet the inclusion criteria will be enrolled in the study and included in the trial. Patients who will not fulfill the inclusion criteria will also be treated but will be excluded from the study analysis.

II-3 Cavity preparation:

The same treatment protocol will be followed for all patients where each patient will receive two compound class II cavities in posterior molar teeth distributed in both sides. Local anesthesia will be administered in the beginning of the session and quadrant isolation will be administrated by rubber dam. Access through enamel and outline form will be obtained with a sterile high speed #245 bur. Following the international guidelines, all soft infected dentine will be removed, and a hard sound dentin floor should be reached. For the peripheries of the cavity, carious tissue removal to hard dentine will be performed using a sharp sterile spoon double-ended excavator and a low-speed round bur. The dentinoenamel junction, cavosurface margins and gingival box will be inspected carefully and to be clean, with at least 1.5 to 2 mm rim of peripheral sound tooth structure to provide a firm marginal adhesion for the restoration.

II-4 Randomization:

To minimize selection bias and ensure equal distribution of treatment protocol across both treated molars, simple randomization will be used to randomly determine which molar receives which material. Therefore, randomization will be performed using an online randomization tool (https://www.randomizer.org/) prior to treatment allocation where, each patient will be given a unique study number, ensuring that each patient receives both treatments in a randomly assigned manner.

II-5 Restorative procedures:

Each included patient with the already prepared cavities will receive two different types of restorations. where one of them will be restored with light cured nano hybrid RBC (Filtek™ Z250, 3M ESPE St.Paul,M,USA) (M1) meanwhile, the second cavity will be restored with self-cure bioactive RBC (Stela, SDI, Australia) (M2).

A sectional matrix system will be used to achieve proper proximal contour and anatomically correct contact with the adjacent tooth. Then, the restorative procedure of each cavity will be carried out according to the manufacturer's recommendations of each tested restoration. Before restoration each cavity will be carefully cleaned with copious air water spray before being dried. Restoration of (M1) group will be performed through selective etching of the prepared cavity enamel surface using 37% phosphoric acid gel (Meta Biomed, Korea) for 15 seconds. This will be followed by rinsing with water for 15 seconds and gentle air drying for 5 seconds, leaving the cavity slightly moist. After that, single layer of a universal adhesive bonding agent (Bisco, INC Schaumburg, IL, USA) will be applied to the prepared cavity walls and floor using disposable adhesive micro brush. The adhesive will be subsequently cured for 20 seconds using LED light curing unit (Elipar S10, 3M ESPE, St Paul, Minnesota, USA) with an intensity of 1200 mW/cm2. The nano hybrid RBC (Filtek™ Z250) will be incrementally applied, and light cured according to manufacturer instructions. Finally, finishing and polishing of the restoration using one-step polishing system (Dimanto, Voco, Germany). Then, checking of occlusion and proximal contacts will be done.

Restoration of (M2) group will be performed through conditioning of cavities with a specialized primer (STELA primer, SDI, Australia) according to manufacturer instructions. Then, a self cured bioactive RBC (STELA, SDI, Australia) will be placed in a single increment and allowed to self-cure according to manufacturer instructions. Then, finishing and polishing of the restoration, checking the occlusion and proximal contacts will be done as mentioned before.

II-6- Evaluation of the wear resistance:

A digital impression will be taken immediately after restoration (T0) using an intraoral scanner (Helios 600 intraoral scanner, Eighteeth, Changzhou, China). To ensure optimal performance and accuracy, the scanner underwent regular calibration before scanning each patient, following the manufacturer's recommendations. During the scanning procedure, the device will be positioned at a 90° angle for the occlusal surface and at 45° angles for both buccal and lingual surfaces. Later on, each restoration will be examined at standardized follow-up periods; six months (T1), twelve months (T2), eighteen months (T3) and twenty-four months (T4). The 3D impressions will be analyzed using a software (Geomagic software, 3D Systems Inc., USA) program and the impressions of each two consultative visits will be superimposed to determine the wear volume loss (mm3).

II-7- Assessment of the bioactivity:

Bioactivity of each examined restoration will be determined by the evaluation of mineral density beneath the tested materials. Immediately after restoration (D0), an image plate digital sensor (Xios XG Supreme, Dentsply Sirona, UK) will be used for transmitting the radiographic image of the selected tooth to the computer. A posterior parallel kit will be used for image standardization. Later, each restoration will be examined at standardized follow-up periods; one month (D1) and three months (D2). The image plate will be inserted at one end of the parallel kit, while the other end was connected to the x-ray cone. All the radiographs will be evaluated for the outcome by a software (ImageJ software, NIH, USA). The assessment of mineral density will be done by the software through performing the following measurements: in each image a line will be drawn along the CEJ to act as a reference, while another parallel line will be drawn at the bottom of the cavity. The distance between both lines will be standardized for each tooth by measuring the length of a vertical line connecting them. The length of the line centralized at the bottom of the cavity will be determined in pixels directly via the previously mentioned software. Such length will be fixed for each sample throughout assessment intervals. Three points on this line (at its start, middle and end) will be determined. The mineral density value at each of these points will be identified by taking the corresponding three readings from the software and recording them to calculate the average value. The mineral density mean value will be calculated from the software

ELIGIBILITY:
Inclusion Criteria:

* Patients with vital two molar teeth with compound class II deep carious lesions.
* Both males and females will be included.
* Patients with good general health.
* Patients with good oral hygiene.
* Co-operative patients.
* Absence of spontaneous pain, mobility or tenderness on percussion.
* Radiographically: no internal or external resorption, no periapical or furcation radiolucency and no widening of the periodontal ligament space.

Exclusion Criteria:

* Patients with systemic disease.
* Patients with severe or chronic periodontitis.
* Patients having allergy to the materials used in this trial.
* Nonfunctioning teeth.
* Teeth with any pathologic pulpal changes.
* Teeth with previous restorations.
* Teeth with surface loss due to non carious lesions.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-11-22 (Actual); Primary Completion 2026-12-02 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of the bioactivity | immediately after restoration (D0) ; one month (D1) and three months (D2)
  Bioactivity of each examined restoration will be determined by the evaluation of mineral density beneath the tested materials. Immediately after restoration (D0), an image plate digital sensor (Xios XG Supreme, Dentsply Sirona, UK) will be used for transmitting the radiographic image of the selected tooth to the computer. Later, each restoration will be examined at standardized follow-up periods. All the radiographs will be evaluated for the outcome by a software (ImageJ software, NIH, USA).
wear resistance | Immediately after restoration, six months (T1), twelve months (T2), eighteen months (T3) and twenty-four months (T4).
  A digital impression will be taken immediately after restoration (T0) using an intraoral scanner (Helios 600 intraoral scanner, Eighteeth, Changzhou, China). To ensure optimal performance and accuracy, the scanner underwent regular calibration before scanning each patient, following the manufacturer's recommendations. During the scanning procedure, the device will be positioned at a 90° angle for the occlusal surface and at 45° angles for both buccal and lingual surfaces. Later on, each restoration will be examined at standardized follow-up periods; six months (T1), twelve months (T2), eighteen months (T3) and twenty-four months (T4). The 3D impressions will be analyzed using a software (Geomagic software, 3D Systems Inc., USA) program and the impressions of each two consultative visits will be superimposed to determine the wear volume loss (mm3)

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal University, Ismailia, Ismalia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
international puplication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: "The IPD will be available beginning 6 months after publication of the main results, and for a period of 5 years thereafter. Data will be de-identified before sharing
Access Criteria: "Qualified researchers can request access to the data by submitting a formal proposal to the Principal Investigator (PI) that describes the research question, required data, and planned analysis. Access will be granted following a review by the study steering committee and execution of a data sharing agreement

REFERENCES:
- [Background] Elderiny HM, Khallaf YS, Akah MM, Hassanein OE. Clinical Evaluation of Bioactive Injectable Resin Composite vs Conventional Nanohybrid Composite in Posterior Restorations: An 18-Month Randomized Controlled Clinical Trial. J Contemp Dent Pract. 2024 Aug 1;25(8):794-802. doi: 10.5005/jp-journals-10024-3737. PMID 39653674

DOCUMENTS (1):
  • Study Protocol (2025-10-07): https://cdn.clinicaltrials.gov/large-docs/86/NCT07262086/Prot_000.pdf